CLINICAL TRIAL: NCT02313194
Title: Enabling Forelimb Function with Agonist Drug and Epidural Stimulation in SCI
Brief Title: Spinal Cord Neuromodulation for Spinal Cord Injury
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Lu, MD, PhD, Associate Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-001416
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cervical Spinal Cord Injury; Tetraparesis; Tetraplegia
MeSH Terms: conditions — Quadriplegia | interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stimulation (Experimental): Determine if epidural stimulation can improve motor function.
  Interventions: Device: Epidural Stimulation; Drug: Buspirone

INTERVENTIONS:
Device: Epidural Stimulation — Determine if epidural stimulation can improve motor function
Drug: Buspirone — Determine if the pharmacological agent in combination with the stimulator can improve motor function.

SUMMARY:
This study is designed to assess the strategy of using spinal cord stimulation to improve the ability to move in spinal cord injured humans.

DETAILED DESCRIPTION:
An epidural stimulation device will be tested to determine if motor function can be improved.

ELIGIBILITY:
Inclusion Criteria:

1. Stable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate hand/arm movement
2. No severe cardiopulmonary diseases such as severe bradycardia, severe autonomic dysreflexia, and/or Chronic Obstructive Pulmonary Disease.
3. No painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore, or infection that might interfere with upper extremity training
4. No clinically significant depression or ongoing drug abuse
5. No current anti-spasticity medication regimen
6. Non-progressive SCI above C5
7. Must not have received botox injections in the prior six months
8. Be unable to grip or move independently
9. Be at least one-year post injury
10. Must be at least 18 years of age
11. Segmental reflexes remain functional below the lesion
12. Female subjects of child-bearing potential must not be pregnant and must be using a medically acceptable method of contraception
13. No current implant(s) of neurostimulators, cardiac pacemakers, defibrillators, shunts, stents, or aneurysm clips, and must have no future exposure to diathermy following implantation
14. No coagulopathy, cardiac risk factors, or other significant medical risk factors for surgery
15. Must not be involved in another clinical trial
16. Must not have disorders or conditions that would require MRI monitoring

Exclusion Criteria:

None as long as inclusion criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-07; Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of arm/hand function | 24 months
  Formal motor testing

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Lu, MD PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States